CLINICAL TRIAL: NCT06671366
Title: Evaluation of Test-retest Correlation in Isokinetic Shoulder Testing
Brief Title: Test-retest Correlation in Isokinetic Shoulder Testing
Acronym: ISO2024
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-A01269-38; 2024-A01269-38 (Other: ANSM)
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-09

CONDITIONS: Isokinetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- External and internal shoulder rotation force (Experimental): shoulder external and internal rotation force objectively using a Cybex dynamometer in a specific position (seated with the arm at 45° abduction and 30° elevation)
  Interventions: Device: external and internal shoulder rotation using a Cybex dynamometer

INTERVENTIONS:
Device: external and internal shoulder rotation using a Cybex dynamometer — Measurement of the reproducibility, in this precise evaluation position, of the results obtained between the different tests carried out 30 minutes apart, and thus the reliability of each measurement in this test.
  measures :
  * Concentric internal rotation 60degrees/sec
  * Concentric external rotation 60 degrees/sec
  * Concentric internal rotation 180 degrees/sec
  * Concentric external rotation 180 degrees/sec
  * Eccentric internal rotation 60degrees/sec
  * Eccentric external rotation 60degrees/sec

SUMMARY:
This study is a prospective, monocentric interventional clinical study in 30 healthy volunteers.

The aim is to objectively assess shoulder external and internal rotation strength using a Cybex dynamometer in a specific position (seated with the arm at 45° abduction and 30° elevation).

The investigator would like here to determine the reproducibility of measurements in this precise evaluation position, but also to determine reference values in healthy subjects.

The results of this study will enable us to improve our management and establish a database for comparison with pathological subjects.

ELIGIBILITY:
Inclusion Criteria:

* Student of the Montpellier School of Physical Therapy
* Adult having received informed information about the study and signed the consent form

Exclusion Criteria:

* Any history of shoulder pathology in the year preceding the tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Correlation between each measurement at peak torque | 1hour
  Correlation between each measurement at peak torque below, and for each arm (12 correlations) in seated position abduction at 45 and 30 degrees anterior elevation.
  * Concentric internal rotation 60degrees/sec
  * Concentric external rotation 60 degrees/sec
  * Concentric internal rotation 180 degrees/sec
  * Concentric external rotation 180 degrees/sec
  * Eccentric internal rotation 60degrees/sec
  * Eccentric external rotation 60degrees/sec
  Evaluation of results using an intraclass correlation coefficient (ICC).

SECONDARY OUTCOMES:
Data in healthy patients | 1hour
  Evaluation of the peak torque of each measurement in healthy patients, have a database.
Establishing the test's external validity | 1hour
  Validated external test :
  1) External validity
  * Differences between dominant arm / weak arm measurements
  * Differences between eccentric and concentric measurements
  * Difference between "test" and "retest" measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique St Jean Sud de France, Saint-Jean-de-Védas, France